CLINICAL TRIAL: NCT00418080
Title: The Role of HER Receptor Family as Indicator of Prognosis and Drug Responsiveness in Locally Advanced Prostate Cancer
Brief Title: Survival Outcomes and Tumor Molecular Profile Following Bicalutamide Neoadjuvant Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of L'Aquila (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BCLT-1236
Record Dates: First submitted 2007-01-03; First posted 2007-01-04 (Estimated); Last update posted 2007-10-08 (Estimated); Status verified 2007-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — bicalutamide

INTERVENTIONS:
Drug: bicalutamide

SUMMARY:
As clinical primary endpoints we assessed whether existed differences in:

1. PSA recurrence rate stratified according to treatment modalities
2. EGFR and HER2/neu overexpression rate stratified according to treatment modalities
3. PSA recurrence rate stratified according to EGFR and HER2/neu overexpression levels.

As secondary clinical endpoints we assessed whether existed differences in:

1. prostate cancer-specific mortality according to treatment modalities
2. prostate cancer-specific mortality stratified according to EGFR and HER2/neu overexpression levels.

For this purpose a post treatment PSA-doubling time of less than 3 months found following PSA recurrence was considered as a surrogate endpoint for prostate cancer-specific mortality Pre-clinical endpoints As pre-clinical endpoint we assessed whether exist differences in efficacy rate of Bicalutamide and Gefitinib treatment in primary tumor cultures stratified for high and low EGFR and HER2/Neu expression levels. The evaluation of efficacy rate of these treatments was documented by comparing the differences of drugs IC50 values among the groups stratified for EGFR and HER2/Neu levels.

ELIGIBILITY:
Inclusion Criteria:

* Patients were eligible if they had histologically confirmed adenocarcinoma of the prostate and the following high-risk features: (1) clinical stage T3a disease with (2) Gleason sum of 7 with a predominant component of 4 (i.e., Gleason 4 + 3 = 7) or (4) Gleason sum of 8, 9 or 10.

Exclusion Criteria:

* Prior hormonal therapy,
* Prior radiation,
* Prior investigational agents,
* Prior malignancy within the last five years or had any other serious medical or psychiatric condition or illness that would not permit the patient to be managed according to the protocol were excluded.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86
Dates: Start 2002-04; Study Completion 2006-12

PRIMARY OUTCOMES:
PSA recurrence rate stratified according to treatment modalities
EGFR and HER2/neu overexpression rate stratified according to treatment modalities
PSA recurrence rate stratified according to EGFR and HER2/neu overexpression levels.

SECONDARY OUTCOMES:
Prostate cancer-specific mortality according to treatment modalities
Prostate cancer-specific mortality stratified according to EGFR and HER2/neu overexpression levels.
For this purpose a post treatment PSA-doubling time of less than 3 months found following PSA recurrence was considered as a surrogate endpoint for prostate cancer-specific mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Luca Gravina, M.D., Principal Investigator — University of L'Aquila
Locations (1):
- University of L'Aquila, L’Aquila, Abruzzo, Italy